CLINICAL TRIAL: NCT07158879
Title: Skin Reactions Related to Thoracic Implantable Chamber Dressings
Acronym: KPAREAC
Status: Recruiting | Type: Observational
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Other Study IDs: DATA240100 KPAREAC
Record Dates: First submitted 2025-07-10; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-06

CONDITIONS: Skin Diseases
Keywords: cancers treated with chemotherapy; skin reaction; dressings
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thoracic catheter port / 1st line chemotherapy: patients treated with chemotherapy (first-line only) using a thoracic implantable catheter chamber

SUMMARY:
Prospective, multicenter cohort of 500 patients newly treated with systemic chemotherapy with CCI. The main objective of this study is to measure the incidence of skin reactions related to thoracic implantable chamber dressings.

DETAILED DESCRIPTION:
The Implantable Catheter Chamber (ICC) has been in use since the 1980s. It enables the administration of nutrition and/or venotoxic and cytotoxic treatment without altering the patient's venous capital. In oncology, CCIs account for over 90% of central venous accesses used in France, i.e. some 160,000 installations per year.

However, the use of this type of central line can also expose patients to the risk of complications such as infection, obstruction and extravasation, which, given the high stakes for patients, have led to the prioritization of work on these subjects.

To date, studies have focused almost exclusively on infectious risks, which are the most frequent and have the greatest impact on patients. This work has led to improvements in professional practices, such as covering with a semi-permeable film to control the appearance of infectious signs.

Other problems have emerged, such as skin reactions linked to semi-permeable films. These are defined by the appearance of one or more of the following criteria:

* Persistent redness at the dressing site;
* Itching;
* Dermabrasion.

However, little has been written on this subject. A 10-day observational survey was carried out in our oncology departments in 2023:

45.5% of inpatients and 14% of day-care patients (dressing left in place for a few days versus a few hours) developed this type of cutaneous reaction.

Given the high prevalence of these reactions, we feel it is important to see whether these results are confirmed in a large cohort of patients, and to investigate whether skin tolerance could be linked to :

* Individual factors (gender, age, immune status, history, etc.);
* The treatments administered and their side effects on the skin;
* The semi-permeable film and how it was applied;
* Duration of application;
* climatic conditions. To answer these questions, which could lead to proposals for adjustments to good practice in oncology, we propose to carry out a multicenter cohort study.

The study of cutaneous tolerance to CCI dressings is poorly documented. However, it represents a major challenge, due to the repetition of application and removal procedures, the sometimes prolonged duration of application, and can be the cause of discomfort and pain, which can sometimes be considerable.

The choice of a second center in the French West Indies will enable us to observe the cutaneous reactions of a wide variety of skin types, and to observe whether there are differences according to heat and hygrometry. This is an interesting choice in a context of climate change and population mixing.

This care research is complementary to the medical research carried out on CCI infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* New chemotherapy patients (1st line of treatment only)
* Thoracic PAC

Exclusion Criteria:

* PICC Line and femoral PAC;
* Patients undergoing treatment with bi-specific antibodies (e.g. tebentafusp);
* Disunion requiring treatment
* Patients treated for hematological cancer;
* Persons deprived of their liberty or under guardianship (including curatorship);
* Adults under court protection;
* Inability to participate in the study for geographical, social or psychological reasons.
* No inclusion of persons covered by articles L. 1121-5 to L. 1121-8 and L. 1122-1-2 of the French Public Health Code (e.g. minors, protected adults, etc.).
* Opposition to data use

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with thoracic CCI treated with chemotherapy in a day hospital ward at the Institut Curie Paris or the Centre Hospitalier de Polynésie Française or the Uturoa Hospital (French Polynesia).
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-12-10 (Estimated); Study Completion 2026-12-10 (Estimated)

PRIMARY OUTCOMES:
Measuring the incidence of skin reactions associated with thoracic implantable chamber dressings | through study completion, an average of 18 months
  Appearance of itching and/or erythema (defined as diffuse or localized congestive redness of the skin) at the dressing site

SECONDARY OUTCOMES:
Identify risk factors for skin reactions to dressings | through study completion, an average of 18 months
  correlation between the onset of skin reactions and the treatments administered
Identify risk factors for skin reactions to dressings | through study completion, an average of 18 months
  Percentage of patients with skin reactions according to the type of dressing used
Identify risk factors for skin reactions to dressings | through study completion, an average of 18 months
  Percentage of patients with skin reactions according to the immune status (polynuclear/monocytic);
Identify risk factors for skin reactions to dressings | through study completion, an average of 18 months
  Percentage of patients with skin reactions according to the duration of application of dressing
Estimate the consequences of these reactions in terms of therapeutic management (implementation of a specific skin treatment, postponement or cancellation of chemotherapy), complications (catheter infection), patient comfort and satisfaction. | through study completion, an average of 18 months
  Evaluation of pain and discomfort experienced by the patient, measured on a numerical scale scale from 0 to 10 (0 = no pain; 10 = very intense pain)
Estimate the consequences of these reactions in terms of therapeutic management (implementation of a specific skin treatment, postponement or cancellation of chemotherapy), complications (catheter infection), patient comfort and satisfaction. | through study completion, an average of 18 months
  Percentage of patients requiring PAC removal
Estimate the consequences of these reactions in terms of therapeutic management (implementation of a specific skin treatment, postponement or cancellation of chemotherapy), complications (catheter infection), patient comfort and satisfaction. | through study completion, an average of 18 months
  Percentage of patients with catheter infection
Estimate the consequences of these reactions in terms of therapeutic management (implementation of a specific skin treatment, postponement or cancellation of chemotherapy), complications (catheter infection), patient comfort and satisfaction. | through study completion, an average of 18 months
  Percentage of patients requiring postponement or cancellation of their chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Betty LIMIER, Principal Investigator — Institut Curie
Locations (3):
- Institut Curie, Paris, France
- French Polynesia (2):
  - Centre Hospitalier de Polynésie Française CHPF, Pirae
  - Hôpital Uturoa, Uturoa